CLINICAL TRIAL: NCT02207998
Title: The Efficacy of the Homoeopathic Complex and Physiotherapy in the Treatment of Chronic Low Back Pain Due to Osteoarthritis
Brief Title: Efficacy of Homoeopathy and Physiotherapy in Chronic Low Back Pain Due to Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Morris 201005532; AEC49-01-2013 (Other: UJohannesburg)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis, physiotherapy, homeopathy, complex
MeSH Terms: conditions — Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homeopathic complex and physiotherapy (Experimental): Homeopathic complex and physiotherapy: (Arnica montana 6CH, Bryonia alba 6CH, Causticum 6CH, Kalmia latifolia 6CH, Rhus toxicodendron 6CH and Calcarea fluoride 6CH) will comprise of 168 tablets; 56 tablets will be issued forth nightly to assess participant's compliance in taking their medicine. Participants will be given instruction to take two tablets, dissolved under the tongue 20 minutes away from meals, twice daily, starting from day one.
  Physiotherapy treatment will consist of lower back classic massage, lumber joint manipulation and the application of a hot pack. Treatment sessions will last for 30 minutes, once every two weeks at the same physiotherapy practice from the same specific and identified physiotherapist.
  Interventions: Drug: Homeopathic complex and physiotherapy
- Placebo and physiotherapy (Placebo Comparator): Placebo and Physiotherapy: Placebo will comprise of 168 unmedicated lactose tablets; 56 tablets will be issued forth nightly to assess participant's compliance in taking their medicine. Participants will be given instruction to take two tablets, dissolved under the tongue 20 minutes away from meals, twice daily, starting from day one.
  Physiotherapy treatment will consist of lower back classic massage, lumber joint manipulation and the application of a hot pack. Treatment sessions will last for 30 minutes, once every two weeks at the same physiotherapy practice from the same specific and identified physiotherapist .
  Interventions: Drug: Placebo and physiotherapy

INTERVENTIONS:
Drug: Homeopathic complex and physiotherapy — Homoeopathic complex (Arnica montana 6CH, Bryonia alba 6CH, Causticum 6CH, Kalmia latifolia 6CH, Rhus toxicodendron 6CH and Calcarea fluoride 6CH) will comprise of medicated lactose tablets.
  Arms: Homeopathic complex and physiotherapy
Drug: Placebo and physiotherapy — Unmedicated lactose tablets. Physiotherapy: lower back classic massage, lumber joint manipulation and the application of a hot pack
  Arms: Placebo and physiotherapy

SUMMARY:
Osteoarthritis (OA) is a chronic arthropathy characterised by disruption and possible loss of joint cartilage along with other joint changes. OA symptoms include progressively developing joint pain provoked or elicited by activity, joint stiffness that lasts for less than 30 minutes on waking and after activity, and occasional joint swelling. It is a common specific mechanical cause of chronic low back pain. Conventional treatment for OA includes physiotherapy treatment and drugs such as paracetamol, non-steroidal anti-Inflammatory drugs (NSAIDs), intra-articular injection of corticosteroids and surgery, however these may have possible side effects. Arnica montana, Bryonia alba, Rhus toxicodendron, Causticum, Kalmia latifolia and Calcarea fluoride are homoeopathic remedies indicated and used in the treatment of OA, however, there is no evidence of studies conducted on a complex made up of these remedies.

The aim of the study is to investigate the efficacy of the homoeopathic complex (Arnica montana 6CH, Bryonia alba 6CH, Causticum 6CH, Kalmia latifolia 6CH, Rhus toxicodendron 6CH and Calcarea fluoride 6CH) and physiotherapy in the treatment of chronic low back pain due to osteoarthritis, using the Oswestry Low Back Pain Disability Questionnaire, range of motion (ROM) measurement using the attraction tape and the visual analogue pain scale (VAS) .

DETAILED DESCRIPTION:
This study is a six week, double-blinded, placebo-controlled study, involving thirty participants, males and females, aged 45-75 years receiving physiotherapy treatment for OA of the lumbar spine at a specific and identified physiotherapist's private practice. A poster advert , placed in the physiotherapist's private practice, with permission , will be used to recruit participants. Individuals who respond to the poster advert will be provided with information pertaining to the study and will be requested to sign a consent form . A screening examination forming part of the inclusion criteria will be conducted by the researcher. Participants meeting the inclusion criteria will be randomly allocated to a treatment or control group; both groups will receive a standard physiotherapy treatment once every two weeks from the physiotherapist. Treatment will consist of lower back classic massage, lumbar joint manipulation, the application of a hot pack and each treatment session will last for 30 minutes. In addition to physiotherapy treatment, participants will be allocated, either a placebo or the homoeopathic complex, with instruction to take two tablets, dissolved under the tongue 20 minutes away from meals, twice daily, starting from day one. This will comprise of 168 tablets, 56 tablets will be issued forth nightly to assess participant's compliance in taking their medicine.

Four consultations will take place at the physiotherapist's private practise. At the first consultation after having divided participants into the treatment and control group, participants will complete the Oswestry Low Back Pain Disability Questionnaire with the researcher's assistance. The researcher will assess the lumbar spine's ROM using the attraction tape measurement. Participants will be provided with 1 copy of the VAS pain scale with spaces to rate their pain every evening for 14 days and 56 tablets. During the second and third consultation, copies of the VAS pain scale will be collected as well as medication containers, to assess participant's compliance in taking their medication. A subjective and physical examination will be conducted, the Oswestry Low Back Pain Disability Questionnaire will be completed and ROM for the lumbar spine will be measured. Participants will receive tablets and copies of the VAS pain scale. On the forth consultation the researcher will conduct the last subjective and physical examination, complete the last Oswestry Low Back Pain Disability Questionnaire and conduct the last ROM measurement using the attraction tape measurement. The last copies of the VAS pain scale and medication containers will be collected.

A subjective and physical examination, Oswestry Low Back Pain Disability Questionnaire, the retraction tape measurement for ROM and the VAS pain scale will be used to collect data and analysed statistically using the Wilcoxon signed test or t-test within groups and t-test (parametric) or Mann-Whitney U (non-parametric) on between groups

ELIGIBILITY:
Inclusion Criteria:

* Must present with symptomatic chronic lower back pain due to OA for more than 3 months and having been diagnosed by a health care practitioner with OA;
* They must have symptoms of OA such as pain and decreased range of motion, on subjective and physical examination and
* Participants must be receiving physiotherapy treatment from a specific and identified physiotherapist

Exclusion Criteria:

* Participants who are receiving any other forms of therapy other than physical therapy (massage and thermotherapy), for example osteopathy, acupuncture, ultrasound or electrotherapy as part of physiotherapy treatment;
* Those presenting with acute lower back pain (with duration of only 3 months or less) and those suffering from chronic lower back pain as a result of disc herniation, compression fracture, lumbar spinal stenosis or spondylolisthesis.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 6 weeks
  The Oswestry Low Back Pain Disability Questionnaire is a standard and validated Questionnaire used in many studies conducted on low back pain. It measures the intensity of pain, how personal care may be affected by pain, how activities such as lifting, walking, standing, sitting and sleeping may be affected by pain. Each section is scored on a six-point scale (0-5) with 0 representing no limitation and 5 representing a maximal limitation. The total score is 50 which is doubled and interpreted as a percentage of the patient-perceived disability (the higher the score, the greater the disability). This will be completed at week 0, and at the end of weeks 2, 4 and 6.

SECONDARY OUTCOMES:
visual analogue pain scale (VAS) | 6 weeks
  The VAS for pain is also an established and validated tool that is used in determining the subjective level of pain in an individual. It can be used to assess how pain changes with treatment. It will be completed once daily from week 0 to week 6.

OTHER OUTCOMES:
range of motion (ROM) | 6 weeks
  Range of motion is assessed using the attraction tape measurement (a standard validated approach) which involves the use of a tape measure, placed directly over the lumbar spine while the patient bends as far as they can. A 0-cm mark is represented by the spinal intersection of a horizontal line drawn between the left and right posterior superior iliac spines. From this point, a second mark is placed 10 cm superior (flexion reference) and a third mark 5 cm inferior (extension reference). Lumbar flexion and extension is measured using this method and it demonstrates test reliability and can differentiate normal from those with "significantly limiting low back pain". ROM will be assessed every two weeks, from week 0 to week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Tebogo Tsele-Tebakang, M.Tech Hom, Study Director — University of Johannesburg; Elizabeth M Solomon, D.Tech Hom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morris M, Pellow J, Solomon EM, Tsele-Tebakang T. Physiotherapy and a Homeopathic Complex for Chronic Low-back Pain Due to Osteoarthritis: A Randomized, Controlled Pilot Study. Altern Ther Health Med. 2016 Jan-Feb;22(1):48-56. PMID 26773321